CLINICAL TRIAL: NCT05147428
Title: D- PRESCRIBE-AD (The Developing a PRogram to Educate and Sensitize Caregivers to Reduce the Inappropriate Prescription Burden in Elderly With Alzheimer's Disease Study)
Brief Title: A Program to Reduce Inappropriate Medications Among Older Adults With Alzheimer's Disease
Acronym: D-PRESCRIBE-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Harvard Pilgrim Health Care (Other); Humana Co.Ltd. (Industry); Elevance Health (Industry); HealthCore, Inc. (Industry)
Responsible Party: Principal Investigator, Jerry Gurwitz, Professor of Medicine, Family Medicine and Community Health, and Population & Quantitative Health Sciences Chief, Division of Geriatric Medicine UMass Chan Medical School and UMass Memorial Medical Center Executive Director, Meyers Health Care Institute, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00023453; 4R33AG069794-02 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: Deprescribing; Dementia; Medication Safety
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The study design will be a prospective, randomized, "open-label" educational intervention trial with three arms: (1) a combined patient/caregiver and provider educational intervention; (2) a provider only educational intervention; and (3) usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient-Provider (Experimental): Both patients and providers will receive educational materials on inappropriate prescribing and deprescribing.
  Interventions: Other: Educational Materials
- Provider Only (Experimental): Only providers will receive educational materials on inappropriate prescribing and deprescribing.
  Interventions: Other: Educational Materials
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Educational Materials — Educational materials on inappropriate prescribing and deprescribing.
  Arms: Patient-Provider; Provider Only

SUMMARY:
Potentially inappropriate prescribing includes the use of medications that may no longer be necessary or that may increase the risk of harm. Inappropriate prescribing can increase the overall symptom burden, and negatively affect health-related quality of life and function. The inappropriate prescription of certain drug categories such as sedative/hypnotics, antipsychotics, and strong anticholinergic agents poses particular risks for older adults, and may be more common among those with Alzheimer's disease and Alzheimer's disease- related dementias (AD/ADRD) due to a higher prevalence of multimorbidity and more frequent prescription of five or more medications. The D-PRESCRIBE-AD (Developing a PRogram to Educate and Sensitize Caregivers to Reduce the Inappropriate Prescription Burden in Elderly with Alzheimer's Disease) study will test a health plan-based intervention using the NIH Collaboratory's Distributed Research Network, which employs the Food and Drug Administration (FDA) Sentinel System infrastructure. The overarching goal of this randomized controlled trial is to assess the effect of a patient/caregiver- centered, multifaceted educational intervention on potentially inappropriate prescribing in patients with AD/ADRD. The research hypothesis is that education on inappropriate prescribing among patients/caregivers and their providers can reduce medication-related morbidity in patients with AD/ADRD and improve medication safety for this vulnerable population. The study population will include community-dwelling patients with AD/ADRD, identified based on diagnoses codes of AD/ADRD or use of a medication for Alzheimer's Disease, who have evidence of potentially inappropriate prescribing the three drug classes above. The trial will evaluate the effect of educational interventions designed to spur patient/caregiver-provider communication about medication safety (versus usual care) on the proportion of patients with inappropriate prescribing, the primary outcome of this study. The trial will be conducted in two large, national health plans.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Diagnosis of AD/ADRD based on a combination of AD/ADRD codes or treatment with a pharmacologic therapy used for AD (e.g., donepezil, rivastigmine, galantamine, and memantine) in the 365 days prior to or on cohort entry date.
2. Evidence of potentially inappropriate prescribing with antipsychotics, sedative-hypnotics, and strong anticholinergics within the past 3 months
3. Age ≥50 years of age as of cohort entry date
4. Continuous medical and pharmacy insurance coverage for at least the prior year

Patient Exclusion Criteria:

1. Evidence of residing in a nursing home or skilled nursing facility or receiving palliative care.
2. Incomplete/missing prescriber ID or incomplete contact information for either patient or prescribing provider.
3. On "do not contact" list

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14442 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — UMass Chan Medical School; UMass Memorial Medical Center; Meyers Health Care Institute
Locations (1):
- Umass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Li X, Cocoros NM, Antonelli MT, Avula R, Crawford SL, Dashevsky I, Fouayzi H, Harkins TP, Mazor KM, Michnick AI, Parlett L, Paullin M, Platt R, Rochon PA, Saphirak C, Si M, Zhou Y, Gurwitz JH. High-Risk Medications in Persons Living With Dementia: A Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1426-1433. doi: 10.1001/jamainternmed.2024.5632. PMID 39432286
- [Derived] Singh S, Cocoros NM, Li X, Mazor KM, Antonelli MT, Parlett L, Paullin M, Harkins TP, Zhou Y, Rochon PA, Platt R, Dashevsky I, Massino C, Saphirak C, Crawford SL, Gurwitz JH. Developing a PRogram to Educate and Sensitize Caregivers to Reduce the Inappropriate Prescription Burden in the Elderly with Alzheimer's Disease (D-PRESCRIBE-AD): Trial protocol and rationale of an open-label pragmatic, prospective randomized controlled trial. PLoS One. 2024 Feb 12;19(2):e0297562. doi: 10.1371/journal.pone.0297562. eCollection 2024. PMID 38346025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with 1 year of health plan coverage who met the following criteria:
  1) AD/ADRD, defined as either presence of International Statistical Classification of Diseases and Related Health Problems, Tenth Revision codes for AD/ADRD associated with 2 different claims or as 2 dispensings for an agent used for AD in the 365 days prior to or on cohort entry; (2) age 50 or older; and (3) a dispensing of any of the 3 targeted drug classes in the 3 months prior to or on cohort entry.
Pre-assignment Details: To address the potential for within-prescriber contamination, only 1 randomly selected eligible patient was randomized per prescribing clinician.
Groups:
- Usual Care: Usual care - no intervention.
Period: Overall Study
Arm/Group | Patient-Provider | Provider Only | Usual Care
Started (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4814 (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4814 (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4814 (N.B., Providers were NOT enrolled and were NOT study subjects.)
Completed (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4286 (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4230 (N.B., Providers were NOT enrolled and were NOT study subjects.) | 4271 (N.B., Providers were NOT enrolled and were NOT study subjects.)
Not Completed | 528 | 584 | 543
Not completed — Removed prior to mailing | 289 | 306 | 270
Not completed — Died or disenrolled during blackout period | 239 | 278 | 273

BASELINE CHARACTERISTICS:
Population: Modified intention to treat cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-Provider | Provider Only | Usual Care | Total
Number analyzed (Participants) | 4,286 | 4,230 | 4,271 | 12787
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 431 | 427 | 428 | 1286
  >=65 years | 3855 | 3803 | 3843 | 11501
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.4 (9.3) | 77.3 (9.4) | 77.2 (9.3) | 77.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2971 | 2860 | 2911 | 8742
  Male | 1315 | 1370 | 1360 | 4045
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4286 | 4230 | 4271 | 12787
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 8 | 9 | 18
  Asian | 32 | 27 | 25 | 84
  Native Hawaiian or Other Pacific Islander | 40 | 31 | 40 | 111
  Black or African American | 451 | 447 | 443 | 1341
  White | 2779 | 2717 | 2761 | 8257
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 983 | 1000 | 993 | 2976
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4286 | 4230 | 4271 | 12787

OUTCOME MEASURES:

1. Primary Outcome: Time to Dispensing of Inappropriate Medication Prescription
Description: The primary outcome will be defined as dispensing of the targeted inappropriate prescription class from day 91 to day 270 during the 6 months observation period following receipt of intervention, or days 91-270.
Time Frame: 6 months
Population: Modified intention to treat cohort.
Measure: Number (95% Confidence Interval); unit: Percentage of Cumulative Incidence
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 4286 | 4230 | 4271
Percentage of Cumulative Incidence | 76.7 [75.45 to 78.0] | 77.9 [76.5 to 79.1] | 77.5 [76.2 to 78.8]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; For the primary analysis, we combined all three targeted medication classes (antipsychotics, sedative/hypnotics, or strong anticholinergics). We calculated Kaplan-Meier curves and performed log-rank testing, and estimated hazard ratios using Cox proportional hazards modeling, censoring at death or disenrollment from the health plan, or at the end of the 6-month study observation period, whichever came first. The index date for the survival analysis was the end of the 3-month blackout period; Test type: Superiority; p = 0.76, Log Rank; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.94 to 1.04]

2. Secondary Outcome: Dose Reduction
Description: Dose reduction was measured as the percentage of patients who achieved a reduction in the patient-specific and medication-specific mean daily dose of the medication targeted for deprescribing of 50% or more during the 6-month study observation period compared with the mean daily dose for the 6-month period immediately preceding the date of mailing of the educational materials. Mean daily dose was calculated using days of supply, dispensed quantity, and unit strength of all dispensings occurring during the 6-month period of interest (either the 6-month study observation period or the 6-month period immediately preceding the date of the mailing).
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
percentage of participants | 25.8 [24.4 to 27.3] | 24.2 [22.8 to 25.6] | 24.8 [23.4 to 26.2]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; Secondary outcomes were analyzed only for those patients who were not censored due to health plan disenrollment or death over the 6-month study observation period (n = 10 424). For analyses of secondary outcomes, we compared the 3 arms using chi-square testing for dichotomous outcomes; Test type: Superiority; p = 0.33, Chi-squared

3. Secondary Outcome: Percentage of Participants With Polypharmacy
Description: Polypharmacy was defined as being dispensed 5 or more unique prescription medications, assessed on the last day of the 6-month study observation period. Polypharmacy was based on medications administered by any route (including topical or ocular medications) and included AD medications and the 3 medication classes targeted for deprescribing. A combination drug was considered a single medication for the purpose of this analysis.
Time Frame: 6 months
Population: Secondary outcomes were analyzed only for those patients who were not censored due to health plan disenrollment or death over the 6-month study observation period (n = 10 424). For analyses of secondary outcomes, we compared the 3 arms using chi-square testing for dichotomous outcomes.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
Percentage of participants | 81.3 [80.0 to 82.6] | 82.3 [81.0 to 83.5] | 82.0 [80.8 to 83.3]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.55, Chi-squared

4. Secondary Outcome: Percentage of Participants With Ambulatory Encounters
Description: We assessed the occurrence of any ambulatory encounter over the 6-month observation period.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
Percentage of participants | 94.2 [93.4 to 94.9] | 93.8 [93.0 to 94.6] | 94.5 [93.7 to 95.2]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.47, Chi-squared

5. Secondary Outcome: Percentage of Participants Who Died
Description: We assessed all-cause inpatient mortality in all study participants (n=12,787) during the 6-month study observation period.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 4286 | 4230 | 4271
Percentage of participants | 1.2 [0.9 to 1.5] | 1.4 [1.1 to 1.8] | 1.2 [0.9 to 1.6]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; Test type: Superiority; p = 0.66, Log Rank

6. Secondary Outcome: Switching Within Classes
Description: Switching of agents within the following targeted drug classes: sedative/ hypnotics, antipsychotics, highly anticholinergic agents.
Time Frame: 6 months
Population: Data were not collected on this measure.
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Emergency Department Encounters
Description: We assessed the occurrence of any emergency department encounters over the 6-month observation period.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
Percentage of participants | 31.7 [30.1 to 33.2] | 33.0 [31.4 to 34.6] | 33.6 [32.1 to 35.2]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.19, Chi-squared

8. Secondary Outcome: Percentage of Participants With Hospitalizations
Description: We assessed the occurrence of any hospitalizations over the 6-month observation period.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
Percentage of participants | 12.0 [10.9 to 13.1] | 12.9 [11.8 to 14.1] | 12.8 [11.7 to 13.9]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.46, Chi-squared

9. Secondary Outcome: Percentage of Participants With Non-acute Institutional Admissions
Description: We assessed the occurrence of any non-acute institutional admissions over the 6-month observation period.
Time Frame: 6 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patient-Provider | Provider Only | Usual Care
Number analyzed (Participants) | 3498 | 3463 | 3463
Percentage of participants | 7.2 [6.3 to 8.1] | 6.9 [6.1 to 7.8] | 6.8 [5.9 to 7.6]
Statistical Analysis 1: Comparison: Patient-Provider vs Provider Only vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.79, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patient-Provider | Provider Only | Usual Care
All-Cause Mortality (participants affected / at risk) | 51/4286 | 59/4230 | 51/4271
Serious Adverse Events (participants affected / at risk) | 0/4286 | 0/4230 | 0/4271
Other Adverse Events (participants affected / at risk) | 0/4286 | 0/4230 | 0/4271

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT05147428/Prot_SAP_000.pdf